CLINICAL TRIAL: NCT04017221
Title: Safety of Sodium-glucose Cotransporter 2 (SGLT2) Inhibitors Among Patients with Type 2 Diabetes: a Multicenter Cohort Study
Brief Title: Safety of Sodium-glucose Cotransporter 2 (SGLT2) Inhibitors Among Patients with Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Canadian Network for Observational Drug Effect Studies, CNODES (Other)
Collaborators: Drug Safety and Effectiveness Network, Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: Q18-09/10/11
Record Dates: First submitted 2019-07-03; First posted 2019-07-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2020-08

CONDITIONS: Diabetes Mellitus, Type 2; Urosepsis; Diabetic Ketoacidosis; Lower Extremity Amputation
Keywords: Sodium-glucose cotransporter 2 inhibitors; Diabetes mellitus, type 2; Urosepsis; Diabetic ketoacidosis; Lower extremity amputation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Ketoacidosis | interventions — Sodium-Glucose Transporter 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Sodium-glucose cotransporter 2 (SGLT2) inhibitors: Current use of a SGLT2 inhibitor alone or in combination with other antidiabetic drugs, excluding DPP-4 inhibitors and insulin.
  Interventions: Drug: Sodium-glucose cotransporter 2 (SGLT2) inhibitors
- Dipeptidyl peptidase-4 (DPP-4) inhibitors: Current use of a DPP-4 inhibitor alone or in combination with other antidiabetic drugs, excluding SGLT2 inhibitors and insulin.
  Interventions: Drug: Dipeptidyl peptidase-4 (DPP-4) inhibitors
- Other treatment combinations: Current use of other antidiabetic drugs, current use of insulin (alone or combination with other antidiabetic drugs), and non-current use of antidiabetic drugs.
  Interventions: Drug: Other treatment combinations

INTERVENTIONS:
Drug: Sodium-glucose cotransporter 2 (SGLT2) inhibitors — Current exposure to SGLT2 will be defined as a prescription for a SGLT2 inhibitor (canagliflozin, dapagliflozin, empagliflozin) alone or in combination with other antidiabetic drugs, excluding DPP-4 inhibitors and insulin.
  Other Names: ATC A10BK
  Groups: Sodium-glucose cotransporter 2 (SGLT2) inhibitors
Drug: Dipeptidyl peptidase-4 (DPP-4) inhibitors — Current exposure to DPP-4 will be defined as a prescription for a DPP-4 inhibitor (alogliptin, linagliptin, saxagliptin, sitagliptin, vildagliptin) alone or in combination with other antidiabetic drugs, excluding SGLT2 inhibitors and insulin.
  Other Names: ATC A10BH
  Groups: Dipeptidyl peptidase-4 (DPP-4) inhibitors
Drug: Other treatment combinations — Current exposure to other treatment combinations will be defined as a prescription of other antidiabetic drugs (metformin, sulfonylureas, thiazolidinediones, GLP-1 receptor agonists, alpha-glucosidase inhibitors, meglitinides, insulin, or combinations of these drugs), current use of insulin (alone or combination with other antidiabetic drugs), and non-current use of antidiabetic drugs.
  Other Names: ATC A10A and A10B (excluding A10BH and A10BK)
  Groups: Other treatment combinations

SUMMARY:
The purpose of this study is to compare the risk of serious adverse events associated with the use of sodium-glucose cotransporter 2 (SGLT2) inhibitors in comparison with the use of dipeptidyl peptidase-4 (DPP-4) inhibitors among patients with type 2 diabetes. More specifically, the investigators will assess the risk of severe urinary tract infection (urosepsis), diabetic ketoacidosis and lower extremity amputation. The investigators hypothesize that the use of SGLT2 inhibitors will be associated with an increased risk of serious adverse events in comparison with the use of DPP-4 inhibitors.

The investigators will carry out separate population-based cohort studies using health care databases in seven Canadian provinces and the United Kingdom. Separate study cohorts will be created for each of the three safety outcomes. The study cohorts will be defined by the initiation of a SGLT2 inhibitor or a DPP-4 inhibitor after SGLT2 inhibitors entered the market. Patients will be followed up until the occurrence of an adverse event. The results from the separate sites will be combined by meta-analysis to provide an overall assessment of the risk of serious adverse events in users of SGLT2 inhibitors in comparison to users of DPP-4 inhibitors.

DETAILED DESCRIPTION:
The objective of this study is to compare the risk of serious adverse events associated with the use of sodium-glucose cotransporter 2 (SGLT2) inhibitors in comparison with the use of dipeptidyl peptidase-4 (DPP-4) inhibitors among patients with type 2 diabetes. More specifically, the investigators will assess the risk of severe urinary tract infection (urosepsis), diabetic ketoacidosis (DKA) and lower extremity amputation.

A common-protocol approach will be used to conduct retrospective cohort studies using administrative health care data from seven Canadian provinces (Alberta, British Columbia, Manitoba, Nova Scotia, Ontario, Quebec, and Saskatchewan) and the United Kingdom (UK) Clinical Practice Research Datalink (CPRD). Briefly, the Canadian databases include population-level data on physician billing, diagnoses and procedures from hospital discharge abstracts, and dispensations for prescription drugs. The data in Ontario will be restricted to patients aged 65 years old and older. The CPRD is a clinical database that is representative of the UK population and contains the records for patients seen at over 680 general practitioner practices in the UK; these data will be linked to the Hospital Episode Statistics (HES) database, which contains in-hospital diagnosis and procedure data.

In each jurisdiction, the investigators will assemble a source population that includes all patients who received an antidiabetic medication (metformin, sulfonylureas, thiazolidinediones, DPP-4 inhibitors, SGLT2 inhibitors, GLP-1 receptor agonists, alpha-glucosidase inhibitors, meglitinides, insulin, or combinations of these drugs) between January 1, 2006 and June 30, 2018 (or the latest date of data availability at each site). From this source population, a study-specific cohort including all new users of SGLT2 inhibitors or DPP-4 inhibitors between January 1, 2013 and June 30, 2018 (or latest date of data availability at each site) will be created for each safety outcome. Specific exclusion criteria will be applied for each study cohort. Study cohort entry date will be defined by the dispensation date (or prescription for CPRD) of the newly prescribed SGLT2 or DPP-4 inhibitor. Patients will be followed until the occurrence of an event (defined below), death, end of health care coverage, or end of the study period, whichever occurs first.

Exposure will be defined using a time-varying exposure definition in which each person-day of follow-up will be classified into one of the following three mutually-exclusive categories: current use of SGLT2 inhibitors, current use of DPP-4 inhibitors, or other treatment combinations. For all categories, exposed person-time will be defined by the prescription duration plus a 30-day grace period. DPP-4 inhibitors will serve as the reference category as both classes are second- to third-line therapy. The outcome of interests include urosepsis, DKA and lower extremity amputation. In the urosepsis specific-study, Fournier's gangrene will be assessed in descriptive analyses as a secondary outcome.

Statistical analyses will be conducted separately for each study-specific cohort. Site-specific rates and corresponding corresponding 95% confidential intervals (CI) of each safety outcomes will be estimated using the Poisson distribution. Time-dependent Cox proportional hazards models with follow-up time as the underlying time axis will be used to estimate adjusted hazard ratios (HR) and corresponding 95% CI of the association between current use of SGLT2 and DPP-4 inhibitor use and urosepsis, DKA, and lower extremity amputation. As secondary analyses, each safety outcome will be stratified by age (≥70 and <70 years), sex and SGLT2 molecule. Sensitivity analyses will be performed to assess the robustness of study results and address some of the study limitations. Site-specific results will be combined by random-effects meta-analysis to provide an overall assessment of the risk of serious adverse events in users of SGLT2 inhibitors in comparison to users of DPP-4 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Patients who newly initiated a SGLT2 inhibitor or DPP-4 inhibitor between January 1, 2013 and June 30, 2018 (or latest date of data availability at each site)

Exclusion Criteria:

* Patients aged less than 18 years at cohort entry date (<66 years in Ontario)
* Patients with less than 365 days of health care coverage prior to cohort entry
* Patients with a hospitalization for urinary tract infection or acute pyelonephritis in the 30 days prior to cohort entry (for urosepsis study cohort only)
* Patients with spinal cord injuries affecting the bladder (for urosepsis study cohort only)
* Patients with long-term urinary catheter use (for urosepsis study cohort only)
* Patients with a hospitalization for DKA in the year prior to cohort entry (for DKA study cohort only)
* Patients with a history of lower extremity amputation at any time prior to cohort entry (for lower extremity amputation study cohort only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In each jurisdiction, the investigators will assemble a source population that includes all patients who received an antidiabetic medication between January 1, 2006 and June 30, 2018. From this source population, a study cohort including all new users of SGLT2 inhibitors or DPP-4 inhibitors between January 1, 2013 and June 30, 2018 will be created for each safety outcome. Specific exclusion criteria will be applied for each study cohort. Study cohort entry date will be defined by the dispensation date (or prescription for CPRD) of the newly prescribed SGLT2 or DPP-4 inhibitor.
Sampling Method: Probability Sample
Enrollment: 1249636 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence rate of urosepsis | Patients will be followed from the date of study cohort entry until hospitalization for urosepsis, death, end of health care coverage, or for up to 64 months, whichever occurs first.
  Urosepsis will be defined as a hospitalization with a diagnosis of acute pyelonephritis or urinary tract infection with a corresponding code for sepsis, using the following ICD-10-CA codes:
  * Acute pyelonephritis (ICD-10-CA: N10) or urinary tract infection (ICD-10-CA: N30.0, N39.0) in combination with;
  * Sepsis (ICD-10-CA: A41.x, R56.2, R57.2).
Incidence rate of diabetic ketoacidosis (DKA) | Patients will be followed from the date of study cohort entry until hospitalization for DKA, death, end of health care coverage, or for up to 64 months, whichever occurs first.
  DKA will be defined as a hospitalization with a primary diagnosis of DKA or visit to the emergency department (in sites where this data is available) using the following ICD-10-CA codes: E11.10, E11.12, E13.10, E13.12.
Incidence rate of lower extremity amputation | Patients will be followed from the date of study cohort entry until occurrence of a lower extremity amputation, death, end of health care coverage, or for up to 64 months, whichever occurs first.
  Lower extremity amputation will be defined by procedure codes recorded in the hospital discharge abstract or the physician claims using the following CCI (Canadian Classification of Health Interventions) codes: 1VC93, 1VG93, 1VQ93, 1WA93, 1WE93, 1WI93, 1WJ93, 1WK93, 1WL93, 1WM93, 1WN93.

SECONDARY OUTCOMES:
Incidence rate of Fournier's gangrene | Patients will be followed from the date of study cohort entry until occurrence of Fournier's gangrene, death, end of health care coverage, or for up to 64 months, whichever occurs first.
  Fournier's gangrene will be defined as an inpatient diagnosis using the following ICD-10-CA codes: N49.3, N76.8, N76.88.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Ernst, MD, MSc, FRCPC, Principal Investigator — Lady Davis Institute for Medical Research, Jewish General Hospital
Locations (1):
- Lady Davis Institute for Medical Research, Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher A, Fralick M, Filion KB, Dell'Aniello S, Douros A, Tremblay E, Shah BR, Ronksley PE, Alessi-Severini S, Hu N, Bugden SC, Ernst P, Lix LM; Canadian Network for Observational Drug Effect Studies (CNODES) Investigators. Sodium-glucose co-transporter-2 inhibitors and the risk of urosepsis: A multi-site, prevalent new-user cohort study. Diabetes Obes Metab. 2020 Sep;22(9):1648-1658. doi: 10.1111/dom.14082. Epub 2020 Jun 4. PMID 32383792
- [Background] Yu OHY, Dell'Aniello S, Shah BR, Brunetti VC, Daigle JM, Fralick M, Douros A, Hu N, Alessi-Severini S, Fisher A, Bugden SC, Ronksley PE, Filion KB, Ernst P, Lix LM; Canadian Network for Observational Drug Effect Studies (CNODES) Investigators. Sodium-Glucose Cotransporter 2 Inhibitors and the Risk of Below-Knee Amputation: A Multicenter Observational Study. Diabetes Care. 2020 Oct;43(10):2444-2452. doi: 10.2337/dc20-0267. Epub 2020 Aug 5. PMID 32759360
- [Background] Douros A, Lix LM, Fralick M, Dell'Aniello S, Shah BR, Ronksley PE, Tremblay E, Hu N, Alessi-Severini S, Fisher A, Bugden SC, Ernst P, Filion KB; Canadian Network for Observational Drug Effect Studies (CNODES) Investigators. Sodium-Glucose Cotransporter-2 Inhibitors and the Risk for Diabetic Ketoacidosis : A Multicenter Cohort Study. Ann Intern Med. 2020 Sep 15;173(6):417-425. doi: 10.7326/M20-0289. Epub 2020 Jul 28. PMID 32716707
- See also: This is the website describing the general functions of the organization, other CNODES projects, and investigator profiles. — http://www.cnodes.ca